CLINICAL TRIAL: NCT06946238
Title: Accelerated Partial Breast Irradiation in One Fraction for Patients With Early-stage Disease and Favorable Histological Subtypes (Breast-1F).
Brief Title: Single-fraction APBI for Early-stage Breast Cancer With Favorable Histological Subtypes (Breast-1F)
Acronym: Breast-1F
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrei Fodor, MD, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Breast-1F
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Accelerated Partial Breast Irradiation; Adjuvant Radiotherapy; Stereotactic Body Radiotherapy; Simultaneous Integrated Boost; Ultrahypofractionated Radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A total of 311 patients are expected to be enrolled in this prospective randomized study. For the sample size calculation, a 90% power and a significance level α = 5% are set. The hypothesis is that the proportion of patients free from Ipsilateral Breast Tumor Recurrence (IBTR) 5 years after the end of treatment will be no less than 97.8%, with a margin of 5%. A total of 148 patients per arm are required, with an additional 5% (15 patients) to compensate for drop-outs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1- Single-fraction APBI (Experimental): Patients in the study (randomized to arm 1) will be treated with a total dose (TD) of 15.5 Gy to the Planning Tumor Volume (PTV) with simultaneous integrated boost (SIB) to a TD of 21 Gy to the tumor bed. For each patient, a stereotactic radiotherapy treatment plan will be created to ensure adequate coverage of the treatment volumes and the tolerability of the Organs At Risk (OAR). Specific, already validated dose-volume constraints will be applied for the evaluation of OARs. The dose-volume histogram (DVH) for the Gross Tumor Volume (GTV), Clinical Target Volume (CTV), PTV, and OAR will be calculated in order to achieve the best optimization in terms of tolerability and efficacy.
  Interventions: Radiation: Adjuvant single-fraction accelerated partial breast irradiation
- Arm 2- Five-fractions APBI (Active Comparator): Patients randomized to arm 2 will be treated according to the standard APBI protocol of our department (Florence protocol), delivering a TD of 30 Gy in 5 fractions to the tumor bed.
  Interventions: Radiation: Adjuvant single-fraction accelerated partial breast irradiation

INTERVENTIONS:
Radiation: Adjuvant single-fraction accelerated partial breast irradiation — Experimental arm (arm 1-single-fraction APBI) patients will be treated to a total dose (TD) of 15.5 Gy to the PTV with a simultaneous integrated boost (SIB) to a TD of 21 Gy to the tumor bed, while arm 2-five-fractions APBI patients with 30 Gy/ 5 fractions to PTV.
  Other Names: Ultrahypofractionated Radiotherapy

SUMMARY:
This is a prospective, randomized, monocentric, non-inferiority interventional clinical study comparing an Accelerated Partial Breast Irradiation (APBI) for the surgical bed of early-stage breast cancer patients with favorable histological subtypes, using stereotactic radiotherapy in a single dose of 15.5 Gy with Simultaneous Integrated Boost (SIB) to 21 Gy (study treatment, delivered in a single fraction) versus multifractionated radiotherapy of 30 Gy in 5 fractions (standard treatment, delivered in 5 fractions).

DETAILED DESCRIPTION:
The project refers to a study on patients with early-stage breast cancer with pathological Tumor stage (pT) from in situ (pTis) to pT2 up to 3 cm in diameter, and pathological/clinical nodal stage p/cN0, and favorable histology (Luminal A and Luminal B human epidermal growth factor receptor 2 (HER2)-negative subtypes), comparing an APBI treatment delivered with stereotactic radiotherapy to the Planning Target Volume (PTV) of the tumor bed of the breast with a total dose (TD) of 15.5 Gy in one fraction, with simultaneous integrated boost (SIB) to a TD of 21 Gy to the Gross Tumor Volume (GTV) represented by tumor bed, versus 30 Gy in 5 consecutive fractions to the PTV of the tumor bed, according to the standard APBI protocol of the department (Florence protocol).

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of breast cancer
2. Patients aged ≥40 years
3. Signed informed consent
4. Stage pTis-T2, up to 3 cm in the greatest diameter
5. Luminal A and Luminal B HER2-negative histological subtypes
6. Negative surgical margins (≥ 0.2 cm)
7. Negative lymph nodes at sentinel lymph node biopsy, or alternatively with imaging tests (Positron Emission Tomography (PET)/Computed Tomography (CT) and/or axillary ultrasound, and/or breast Magnetic Resonance Imaging (MRI) with and without contrast), or, in rare cases, where still performed, with axillary dissection
8. Clinical M0 (PET/CT and/or bone scintigraphy and/or abdomen-pelvis CT with and without contrast in suspected patients), within the previous 3 months.
9. Performance Status (PS) Eastern Cooperative Oncology Group (ECOG) ≤2
10. No prior thoracic radiotherapy
11. Fertile women using contraception methods initiated during oncological treatment.

Exclusion Criteria:

1. Patients aged < 40 years
2. Tumors > 3 cm
3. Multicentric tumors
4. Positive or close surgical margins (<0.2 cm)
5. Lobular carcinoma
6. Negative hormone receptors
7. HER2-positive
8. BReast CAncer (BRCA) genes BRCA1 and/or BRCA2 positive (only if known)
9. Severe systemic diseases
10. Psychiatric or other disorders that may prevent the patient from signing informed consent
11. Previous invasive cancer, except for skin cancer (excluding melanoma) unless the patient has been disease-free for at least 3 years (e.g., carcinoma in situ of the oral cavity or bladder)
12. Collagen or autoimmune diseases (systemic lupus erythematosus, rheumatoid arthritis, scleroderma, Sjogren's syndrome)
13. Lymph node disease (N1)
14. Evidence of distant metastasis (M1)
15. Contraindication to systemic treatment
16. Pregnant women
17. Non-compliance with the dose limits established in the treatment plan

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients aged ≥40 years, with early-stage breast cancer and favorable histology will be enrolled
Enrollment: 311 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2035-06-30 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral Breast Tumor Recurrence (IBTR) | 5 years
  To demonstrate the non-inferiority of local control (ipsilateral breast tumor recurrence - IBTR) of the study treatment (delivered in a single-fraction APBI) compared to the department's standard APBI treatment (delivered in 5 fractions).

SECONDARY OUTCOMES:
Acute toxicity | 1 month
  Acute toxicity grade ≥3 as the maximum toxicity value within 1 month and 3 months after the completion of radiotherapy treatment evaluated with Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC) scale with 4 grades, from 0 no change to 4, worst toxicity
Acute toxicity | 3 months
  Acute toxicity grade ≥3 as the maximum toxicity value within 1 month and 3 months after the completion of radiotherapy treatment evaluated with RTOG/EORTC scale with 4 grades, from 0 no change to 4, worst toxicity
Late toxicity | 5 years
  Late toxicity evaluated with RTOG/EORTC and Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, with 5 grades, from 0 = no change, to 5 = death for toxicity
Local Control | 5 years
  Local control of the treated site expressed in terms of local recurrence rate
Local Relapse-Free Survival (LRFS) | From the date of radiotherapy end until the date of local relapse, assessed up to 5 years
  Time to local recurrence
Regional Relapse-Free Survival (RRFS) | From the date of radiotherapy end until the date of regional relapse, assessed up to 5 years
  Time to regional (nodal) recurrence
Distant Metastasis-Free Survival (DMFS) | From the date of radiotherapy end until the date of distant metasis diagnosis, assessed up to 5 years
  Time to distant (metastatic) relapse
Disease-Free Survival (DFS) | From the date of radiotherapy end until the date of first, any ( local, regional, distant) relapse, assessed up to 5 years
  Time to first any relapse: local, regional or distant
Breast Cancer Specific Survival (BCSS) | From the date of radiotherapy end until the date of death from breast cancer, assessed up to 5 years
  Time until death from breast cancer
Overall Survival (OS) | From the date of radiotherapy end until the date of death from any cause, assessed up to 5 years
  Time until death from any cause
Cosmesis | 5 years
  Cosmetic results evaluated with Harvard scale. It assesses the global esthetic appearance of the breast, categorized as Excellent, Good, Fair, or Poor
Acute toxicity interim analysis | 3 months
  An interim analysis of acute toxicity (with RTOG/EORTC andf CTCAE v5.0 scales) will be performed for the first 120 patients
Late toxicity interim analysis | 42 months
  An interim analysis of late toxicity (with RTOG/EORTC andf CTCAE v5.0 scales) will be performed for the first 120 patients
Local relapse interim analysis | 42 months
  An interim analysis of local relapse rate will be performed for the first 120 patients

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed with breast tumor specific quality of life questionnaires | 5 years
  Survey with the questionnaire of European Organisation for Research and Treatment of Cancer (EORTC) Quality of life of brain tumor patients (EORTC QLQ BR42) which contains 42 questions on patients' quality of life with answers from 1, lowest grade, to 4, highest grade
Modeling of organ movement | 5 days
  Modeling of organ movement during treatment
Radiomics | 5 years
  Evaluation of radiomic characteristics: Mathematical extraction of the spatial distribution of signal intensities and pixel interrelationships of medical images of the patients, to quantify textural information resampled according to International Biomarker Standardization Initiative (IBSI).
Predictive factors for toxicity, disease progression and death | 5 years
  Identification of clinical, imaging, and laboratory prognostic factors for an aggressive phenotype of Luminal A and Luminal B HER2-negative breast cancer and for toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Fodor, MD, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study (anonymized individual participant data) are available on request from the corresponding author to researchers who provide a methodologically sound proposal. Requests made to the corresponding author will be evaluated by the Lombardy Territorial Ethics Committee 1
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: for 5 years after the end of the study
Access Criteria: request from the corresponding author approved by the Lombardy Territorial Ethics Committee

REFERENCES:
- [Result] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Result] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Result] Litiere S, Werutsky G, Fentiman IS, Rutgers E, Christiaens MR, Van Limbergen E, Baaijens MH, Bogaerts J, Bartelink H. Breast conserving therapy versus mastectomy for stage I-II breast cancer: 20 year follow-up of the EORTC 10801 phase 3 randomised trial. Lancet Oncol. 2012 Apr;13(4):412-9. doi: 10.1016/S1470-2045(12)70042-6. Epub 2012 Feb 27. PMID 22373563
- [Result] Romestaing P, Lehingue Y, Carrie C, Coquard R, Montbarbon X, Ardiet JM, Mamelle N, Gerard JP. Role of a 10-Gy boost in the conservative treatment of early breast cancer: results of a randomized clinical trial in Lyon, France. J Clin Oncol. 1997 Mar;15(3):963-8. doi: 10.1200/JCO.1997.15.3.963. PMID 9060534
- [Result] Bartelink H, Horiot JC, Poortmans PM, Struikmans H, Van den Bogaert W, Fourquet A, Jager JJ, Hoogenraad WJ, Oei SB, Warlam-Rodenhuis CC, Pierart M, Collette L. Impact of a higher radiation dose on local control and survival in breast-conserving therapy of early breast cancer: 10-year results of the randomized boost versus no boost EORTC 22881-10882 trial. J Clin Oncol. 2007 Aug 1;25(22):3259-65. doi: 10.1200/JCO.2007.11.4991. Epub 2007 Jun 18. PMID 17577015
- [Result] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Result] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bentzen SM, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial B of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet. 2008 Mar 29;371(9618):1098-107. doi: 10.1016/S0140-6736(08)60348-7. Epub 2008 Mar 19. PMID 18355913
- [Result] Whelan T, MacKenzie R, Julian J, Levine M, Shelley W, Grimard L, Lada B, Lukka H, Perera F, Fyles A, Laukkanen E, Gulavita S, Benk V, Szechtman B. Randomized trial of breast irradiation schedules after lumpectomy for women with lymph node-negative breast cancer. J Natl Cancer Inst. 2002 Aug 7;94(15):1143-50. doi: 10.1093/jnci/94.15.1143. PMID 12165639
- [Result] Strnad V, Ott OJ, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Dunst J, Gutierrez Miguelez C, Slampa P, Allgauer M, Lossl K, Polat B, Kovacs G, Fischedick AR, Wendt TG, Fietkau R, Hindemith M, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Schlamann A, Potter R, Gall C, Malzer M, Uter W, Polgar C; Groupe Europeen de Curietherapie of European Society for Radiotherapy and Oncology (GEC-ESTRO). 5-year results of accelerated partial breast irradiation using sole interstitial multicatheter brachytherapy versus whole-breast irradiation with boost after breast-conserving surgery for low-risk invasive and in-situ carcinoma of the female breast: a randomised, phase 3, non-inferiority trial. Lancet. 2016 Jan 16;387(10015):229-38. doi: 10.1016/S0140-6736(15)00471-7. Epub 2015 Oct 19. PMID 26494415
- [Result] Vicini FA, Cecchini RS, White JR, Arthur DW, Julian TB, Rabinovitch RA, Kuske RR, Ganz PA, Parda DS, Scheier MF, Winter KA, Paik S, Kuerer HM, Vallow LA, Pierce LJ, Mamounas EP, McCormick B, Costantino JP, Bear HD, Germain I, Gustafson G, Grossheim L, Petersen IA, Hudes RS, Curran WJ Jr, Bryant JL, Wolmark N. Long-term primary results of accelerated partial breast irradiation after breast-conserving surgery for early-stage breast cancer: a randomised, phase 3, equivalence trial. Lancet. 2019 Dec 14;394(10215):2155-2164. doi: 10.1016/S0140-6736(19)32514-0. Epub 2019 Dec 5. PMID 31813636
- [Result] Whelan TJ, Julian JA, Berrang TS, Kim DH, Germain I, Nichol AM, Akra M, Lavertu S, Germain F, Fyles A, Trotter T, Perera FE, Balkwill S, Chafe S, McGowan T, Muanza T, Beckham WA, Chua BH, Gu CS, Levine MN, Olivotto IA; RAPID Trial Investigators. External beam accelerated partial breast irradiation versus whole breast irradiation after breast conserving surgery in women with ductal carcinoma in situ and node-negative breast cancer (RAPID): a randomised controlled trial. Lancet. 2019 Dec 14;394(10215):2165-2172. doi: 10.1016/S0140-6736(19)32515-2. Epub 2019 Dec 5. PMID 31813635
- [Result] Coles CE, Griffin CL, Kirby AM, Titley J, Agrawal RK, Alhasso A, Bhattacharya IS, Brunt AM, Ciurlionis L, Chan C, Donovan EM, Emson MA, Harnett AN, Haviland JS, Hopwood P, Jefford ML, Kaggwa R, Sawyer EJ, Syndikus I, Tsang YM, Wheatley DA, Wilcox M, Yarnold JR, Bliss JM; IMPORT Trialists. Partial-breast radiotherapy after breast conservation surgery for patients with early breast cancer (UK IMPORT LOW trial): 5-year results from a multicentre, randomised, controlled, phase 3, non-inferiority trial. Lancet. 2017 Sep 9;390(10099):1048-1060. doi: 10.1016/S0140-6736(17)31145-5. Epub 2017 Aug 2. PMID 28779963
- [Result] Meattini I, Marrazzo L, Saieva C, Desideri I, Scotti V, Simontacchi G, Bonomo P, Greto D, Mangoni M, Scoccianti S, Lucidi S, Paoletti L, Fambrini M, Bernini M, Sanchez L, Orzalesi L, Nori J, Bianchi S, Pallotta S, Livi L. Accelerated Partial-Breast Irradiation Compared With Whole-Breast Irradiation for Early Breast Cancer: Long-Term Results of the Randomized Phase III APBI-IMRT-Florence Trial. J Clin Oncol. 2020 Dec 10;38(35):4175-4183. doi: 10.1200/JCO.20.00650. Epub 2020 Aug 24. PMID 32840419
- [Result] Meduri B, Baldissera A, Iotti C, Scheijmans LJEE, Stam MR, Parisi S, Boersma LJ, Ammendolia I, Koiter E, Valli M, Scandolaro L, Busz D, Stenfert Kroese MC, Ciabatti S, Giacobazzi P, Ruggieri MP, Engelen A, Munafo T, Westenberg AH, Verhoeven K, Vicini R, D'Amico R, Lohr F, Bertoni F, Poortmans P, Frezza GP. Cosmetic Results and Side Effects of Accelerated Partial-Breast Irradiation Versus Whole-Breast Irradiation for Low-Risk Invasive Carcinoma of the Breast: The Randomized Phase III IRMA Trial. J Clin Oncol. 2023 Apr 20;41(12):2201-2210. doi: 10.1200/JCO.22.01485. Epub 2023 Jan 9. PMID 36623246
- [Result] Bhattacharya IS, Haviland JS, Kirby AM, Kirwan CC, Hopwood P, Yarnold JR, Bliss JM, Coles CE; IMPORT Trialists. Patient-Reported Outcomes Over 5 Years After Whole- or Partial-Breast Radiotherapy: Longitudinal Analysis of the IMPORT LOW (CRUK/06/003) Phase III Randomized Controlled Trial. J Clin Oncol. 2019 Feb 1;37(4):305-317. doi: 10.1200/JCO.18.00982. Epub 2018 Dec 11. PMID 30532984
- [Result] Benda RK, Yasuda G, Sethi A, Gabram SG, Hinerman RW, Mendenhall NP. Breast boost: are we missing the target? Cancer. 2003 Feb 15;97(4):905-9. doi: 10.1002/cncr.11142. PMID 12569589
- [Result] Vaidya JS, Tobias JS, Baum M, Keshtgar M, Joseph D, Wenz F, Houghton J, Saunders C, Corica T, D'Souza D, Sainsbury R, Massarut S, Taylor I, Hilaris B. Intraoperative radiotherapy for breast cancer. Lancet Oncol. 2004 Mar;5(3):165-73. doi: 10.1016/S1470-2045(04)01412-3. PMID 15003199
- [Result] Vaidya JS, Wenz F, Bulsara M, Tobias JS, Joseph DJ, Keshtgar M, Flyger HL, Massarut S, Alvarado M, Saunders C, Eiermann W, Metaxas M, Sperk E, Sutterlin M, Brown D, Esserman L, Roncadin M, Thompson A, Dewar JA, Holtveg HM, Pigorsch S, Falzon M, Harris E, Matthews A, Brew-Graves C, Potyka I, Corica T, Williams NR, Baum M; TARGIT trialists' group. Risk-adapted targeted intraoperative radiotherapy versus whole-breast radiotherapy for breast cancer: 5-year results for local control and overall survival from the TARGIT-A randomised trial. Lancet. 2014 Feb 15;383(9917):603-13. doi: 10.1016/S0140-6736(13)61950-9. Epub 2013 Nov 11. PMID 24224997
- [Result] Veronesi U, Orecchia R, Maisonneuve P, Viale G, Rotmensz N, Sangalli C, Luini A, Veronesi P, Galimberti V, Zurrida S, Leonardi MC, Lazzari R, Cattani F, Gentilini O, Intra M, Caldarella P, Ballardini B. Intraoperative radiotherapy versus external radiotherapy for early breast cancer (ELIOT): a randomised controlled equivalence trial. Lancet Oncol. 2013 Dec;14(13):1269-77. doi: 10.1016/S1470-2045(13)70497-2. Epub 2013 Nov 11. PMID 24225155
- [Result] Stroom J, Schlief A, Alderliesten T, Peterse H, Bartelink H, Gilhuijs K. Using histopathology breast cancer data to reduce clinical target volume margins at radiotherapy. Int J Radiat Oncol Biol Phys. 2009 Jul 1;74(3):898-905. doi: 10.1016/j.ijrobp.2009.01.026. Epub 2009 May 4. PMID 19409724
- [Result] Darby SC, Ewertz M, McGale P, Bennet AM, Blom-Goldman U, Bronnum D, Correa C, Cutter D, Gagliardi G, Gigante B, Jensen MB, Nisbet A, Peto R, Rahimi K, Taylor C, Hall P. Risk of ischemic heart disease in women after radiotherapy for breast cancer. N Engl J Med. 2013 Mar 14;368(11):987-98. doi: 10.1056/NEJMoa1209825. PMID 23484825
- [Result] Hepel JT, Wazer DE. Partial Breast Irradiation Is the Preferred Standard of Care for a Majority of Women With Early-Stage Breast Cancer. J Clin Oncol. 2020 Jul 10;38(20):2268-2272. doi: 10.1200/JCO.19.02594. Epub 2020 May 22. No abstract available. PMID 32442074
- [Result] Fodor A, Brombin C, Mangili P, Borroni F, Pasetti M, Tummineri R, Zerbetto F, Longobardi B, Perna L, Dell'Oca I, Deantoni CL, Deli AM, Chiara A, Broggi S, Castriconi R, Esposito PG, Slim N, Passoni P, Baroni S, Villa SL, Rancoita PMV, Fiorino C, Del Vecchio A, Bianchini G, Gentilini OD, Di Serio MS, Di Muzio NG. Impact of molecular subtype on 1325 early-stage breast cancer patients homogeneously treated with hypofractionated radiotherapy without boost: Should the indications for radiotherapy be more personalized? Breast. 2021 Feb;55:45-54. doi: 10.1016/j.breast.2020.12.004. Epub 2020 Dec 9. PMID 33326894
- [Result] Bane AL, Whelan TJ, Pond GR, Parpia S, Gohla G, Fyles AW, Pignol JP, Pritchard KI, Chambers S, Levine MN. Tumor factors predictive of response to hypofractionated radiotherapy in a randomized trial following breast conserving therapy. Ann Oncol. 2014 May;25(5):992-8. doi: 10.1093/annonc/mdu090. Epub 2014 Feb 20. PMID 24562444
- [Result] Goldhirsch A, Gelber RD, Piccart-Gebhart MJ, de Azambuja E, Procter M, Suter TM, Jackisch C, Cameron D, Weber HA, Heinzmann D, Dal Lago L, McFadden E, Dowsett M, Untch M, Gianni L, Bell R, Kohne CH, Vindevoghel A, Andersson M, Brunt AM, Otero-Reyes D, Song S, Smith I, Leyland-Jones B, Baselga J; Herceptin Adjuvant (HERA) Trial Study Team. 2 years versus 1 year of adjuvant trastuzumab for HER2-positive breast cancer (HERA): an open-label, randomised controlled trial. Lancet. 2013 Sep 21;382(9897):1021-8. doi: 10.1016/S0140-6736(13)61094-6. Epub 2013 Jul 18. PMID 23871490
- [Result] Fodor A, Brombin C, Mangili P, Tummineri R, Pasetti M, Zerbetto F, Longobardi B, Galvan AS, Deantoni CL, Dell'Oca I, Castriconi R, Esposito PG, Deli AM, Rancoita PMV, Fiorino C, Vecchio AD, Di Serio MS, Di Muzio NG. Toxicity of Hypofractionated Whole Breast Radiotherapy Without Boost and Timescale of Late Skin Responses in a Large Cohort of Early-Stage Breast Cancer Patients. Clin Breast Cancer. 2022 Jun;22(4):e480-e487. doi: 10.1016/j.clbc.2021.11.008. Epub 2021 Dec 1. PMID 34955430
- [Result] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Result] Meattini I, Francolini G, Di Cataldo V, Visani L, Becherini C, Scoccimarro E, Salvestrini V, Bellini C, Masi L, Doro R, Di Naro F, Loi M, Salvatore G, Simontacchi G, Greto D, Bernini M, Nori J, Orzalesi L, Bianchi S, Mangoni M, Livi L. Preoperative robotic radiosurgery for early breast cancer: Results of the phase II ROCK trial (NCT03520894). Clin Transl Radiat Oncol. 2022 Sep 22;37:94-100. doi: 10.1016/j.ctro.2022.09.004. eCollection 2022 Nov. PMID 36177053
- [Result] Zerella MA, Zaffaroni M, Ronci G, Dicuonzo S, Rojas DP, Morra A, Fodor C, Rondi E, Vigorito S, Botta F, Cremonesi M, Garibaldi C, Penco S, Galimberti VE, Intra M, Gandini S, Barberis M, Renne G, Cattani F, Veronesi P, Orecchia R, Jereczek-Fossa BA, Leonardi MC. Single fraction ablative preoperative radiation treatment for early-stage breast cancer: the CRYSTAL study - a phase I/II clinical trial protocol. BMC Cancer. 2022 Apr 2;22(1):358. doi: 10.1186/s12885-022-09305-w. PMID 35366825
- [Result] Murray Brunt A, Haviland JS, Wheatley DA, Sydenham MA, Alhasso A, Bloomfield DJ, Chan C, Churn M, Cleator S, Coles CE, Goodman A, Harnett A, Hopwood P, Kirby AM, Kirwan CC, Morris C, Nabi Z, Sawyer E, Somaiah N, Stones L, Syndikus I, Bliss JM, Yarnold JR; FAST-Forward Trial Management Group. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial. Lancet. 2020 May 23;395(10237):1613-1626. doi: 10.1016/S0140-6736(20)30932-6. Epub 2020 Apr 28. PMID 32580883
- [Result] Civil YA, Vasmel JE, Charaghvandi RK, Houweling AC, Vreuls CPH, van Diest PJ, Witkamp AJ, Doeksen A, van Dalen T, Felderhof J, van Dam I, Slotman BJ, Kirby AM, Verkooijen HM, van der Velde S, van der Leij F, van den Bongard HJGD. Preoperative Magnetic Resonance Guided Single-Dose Partial Breast Irradiation: 5-Year Results of the Prospective Single-Arm ABLATIVE Trial. Int J Radiat Oncol Biol Phys. 2025 Mar 1;121(3):613-622. doi: 10.1016/j.ijrobp.2024.07.2326. Epub 2024 Aug 2. PMID 39098432
- [Result] Bosma SCJ, Leij F, Vreeswijk S, Maaker M, Wesseling J, Vijver MV, Scholten A, Rivera S, Bourgier C, Auzac G, Foukakis T, Lekberg T, Bongard D, Loo C, Rutgers E, Bartelink H, Elkhuizen PHM. Five-Year Results of the Preoperative Accelerated Partial Breast Irradiation (PAPBI) Trial. Int J Radiat Oncol Biol Phys. 2020 Apr 1;106(5):958-967. doi: 10.1016/j.ijrobp.2019.12.037. Epub 2020 Jan 25. PMID 31987957
- [Result] van der Leij F, Bosma SC, van de Vijver MJ, Wesseling J, Vreeswijk S, Rivera S, Bourgier C, Garbay JR, Foukakis T, Lekberg T, van den Bongard DH, van Vliet-Vroegindeweij C, Bartelink H, Rutgers EJ, Elkhuizen PH. First results of the preoperative accelerated partial breast irradiation (PAPBI) trial. Radiother Oncol. 2015 Mar;114(3):322-7. doi: 10.1016/j.radonc.2015.02.002. Epub 2015 Feb 17. PMID 25701298
- [Result] Whelan TJ, Kim DH, Sussman J. Clinical experience using hypofractionated radiation schedules in breast cancer. Semin Radiat Oncol. 2008 Oct;18(4):257-64. doi: 10.1016/j.semradonc.2008.04.008. PMID 18725113
- [Result] Qi XS, White J, Li XA. Is alpha/beta for breast cancer really low? Radiother Oncol. 2011 Aug;100(2):282-8. doi: 10.1016/j.radonc.2011.01.010. Epub 2011 Feb 28. PMID 21367477
- [Result] Ray KJ, Sibson NR, Kiltie AE. Treatment of Breast and Prostate Cancer by Hypofractionated Radiotherapy: Potential Risks and Benefits. Clin Oncol (R Coll Radiol). 2015 Jul;27(7):420-6. doi: 10.1016/j.clon.2015.02.008. Epub 2015 Mar 7. PMID 25752244
- [Result] Brand DH, Kirby AM, Yarnold JR, Somaiah N. How Low Can You Go? The Radiobiology of Hypofractionation. Clin Oncol (R Coll Radiol). 2022 May;34(5):280-287. doi: 10.1016/j.clon.2022.02.009. Epub 2022 Mar 5. PMID 35260319
- [Result] van Leeuwen CM, Oei AL, Crezee J, Bel A, Franken NAP, Stalpers LJA, Kok HP. The alfa and beta of tumours: a review of parameters of the linear-quadratic model, derived from clinical radiotherapy studies. Radiat Oncol. 2018 May 16;13(1):96. doi: 10.1186/s13014-018-1040-z. PMID 29769103
- [Result] Brown JM, Carlson DJ, Brenner DJ. The tumor radiobiology of SRS and SBRT: are more than the 5 Rs involved? Int J Radiat Oncol Biol Phys. 2014 Feb 1;88(2):254-62. doi: 10.1016/j.ijrobp.2013.07.022. PMID 24411596
- [Result] Guidolin K, Yaremko B, Lynn K, Gaede S, Kornecki A, Muscedere G, BenNachum I, Shmuilovich O, Mouawad M, Yu E, Sexton T, Gelman N, Moiseenko V, Brackstone M, Lock M. Stereotactic image-guided neoadjuvant ablative single-dose radiation, then lumpectomy, for early breast cancer: the SIGNAL prospective single-arm trial of single-dose radiation therapy. Curr Oncol. 2019 Jun;26(3):e334-e340. doi: 10.3747/co.26.4479. Epub 2019 Jun 1. PMID 31285677
- [Result] Major T, Gutierrez C, Guix B, van Limbergen E, Strnad V, Polgar C; Breast Cancer Working Group of GEC-ESTRO. Recommendations from GEC ESTRO Breast Cancer Working Group (II): Target definition and target delineation for accelerated or boost partial breast irradiation using multicatheter interstitial brachytherapy after breast conserving open cavity surgery. Radiother Oncol. 2016 Jan;118(1):199-204. doi: 10.1016/j.radonc.2015.12.006. Epub 2016 Jan 8. PMID 26776444
- [Result] Chiappa C, Rovera F, Corben AD, Fachinetti A, De Berardinis V, Marchionini V, Rausei S, Boni L, Dionigi G, Dionigi R. Surgical margins in breast conservation. Int J Surg. 2013;11 Suppl 1:S69-72. doi: 10.1016/S1743-9191(13)60021-7. PMID 24380558
- [Result] Pilewskie M, Morrow M. Margins in breast cancer: How much is enough? Cancer. 2018 Apr 1;124(7):1335-1341. doi: 10.1002/cncr.31221. Epub 2018 Jan 16. PMID 29338088
- [Result] Duane F, Aznar MC, Bartlett F, Cutter DJ, Darby SC, Jagsi R, Lorenzen EL, McArdle O, McGale P, Myerson S, Rahimi K, Vivekanandan S, Warren S, Taylor CW. A cardiac contouring atlas for radiotherapy. Radiother Oncol. 2017 Mar;122(3):416-422. doi: 10.1016/j.radonc.2017.01.008. Epub 2017 Feb 21. PMID 28233564
- [Result] Lozza L, Fariselli L, Sandri M, Rampa M, Pinzi V, De Santis MC, Franceschini M, Trecate G, Maugeri I, Fumagalli L, Bonfantini F, Bianchi G, Pignoli E, De Martin E, Agresti R. Partial breast irradiation with CyberKnife after breast conserving surgery: a pilot study in early breast cancer. Radiat Oncol. 2018 Mar 23;13(1):49. doi: 10.1186/s13014-018-0991-4. PMID 29566762
- [Result] Kennedy WR, Thomas MA, Stanley JA, Luo J, Ochoa LL, Clifton KK, Cyr AE, Margenthaler JA, DeWees TA, Price A, Kashani R, Green O, Zoberi I. Single-Institution Phase 1/2 Prospective Clinical Trial of Single-Fraction, High-Gradient Adjuvant Partial-Breast Irradiation for Hormone Sensitive Stage 0-I Breast Cancer. Int J Radiat Oncol Biol Phys. 2020 Jun 1;107(2):344-352. doi: 10.1016/j.ijrobp.2020.02.021. Epub 2020 Feb 19. PMID 32084524